CLINICAL TRIAL: NCT01172028
Title: Phase I Dose Escalation Trial of Biweekly Alimta (With Vitamin Supplementation) in Combination With Taxotere in Advanced Solid Tumor Patients
Brief Title: Pemetrexed Disodium and Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0108-04; P30CA023074 (NIH); UARIZ-05-0108-01 (Other: University of Arizona); UARIZ-HSC0529 (Other: University of Arizona); UARIZ-SRC17855 (Other: University of Arizona); LILLY-UARIZ-05-0108-01 (Other: University of Arizona)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer; Esophageal Cancer; Gastric Cancer; Head and Neck Cancer; Lung Cancer; Ovarian Cancer; Prostate Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; male breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent lymphoepithelioma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent hypopharyngeal cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent laryngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer
MeSH Terms: conditions — Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms, Male; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Carcinoma, Ovarian Epithelial; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alimta and Taxotere (Experimental): Alimta and Taxotere given in combination with dose modifications.
  Interventions: Drug: Taxotere (Docetaxel); Drug: Alimta (Pemetrexed)

INTERVENTIONS:
Drug: Taxotere (Docetaxel) — Taxotere is a third generation cytotoxic chemotherapy agent which is a semisynthetic taxane that inhibits cell division by promoting the rate of microtubule assembly and preventing microtubule depolymerization. It has broad antitumor activity in a range of solid tumors, and has been studied on a weekly as well as a biweekly dosing schedule.
  Other Names: Docetaxel
Drug: Alimta (Pemetrexed) — ALIMTA is a novel antifolate drug with three enzyme targets in the purine and pyrimidine synthetic pathway. It has broad activity in solid tumors and has been combined with a number of other chemotherapy agents. Its toxicity is modified by the use of continuous vitamin supplementation.
  Other Names: Pemetrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells of by stopping them from dividing. Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of giving pemetrexed disodium and docetaxel together in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of the combination of pemetrexed disodium and docetaxel when administered on a day 1 and day 15 dosing schedule.

Secondary

* To specifically characterize the toxicity profile for the combination of biweekly pemetrexed disodium and docetaxel.
* To investigate the antitumor activity in patients with advanced solid tumors as measured by RECIST criteria for patients with measurable disease or tumor markers for patients with non-measurable disease.
* To determine the recommended phase II dose of the combination of pemetrexed disodium and docetaxel on a biweekly dosing schedule.

OUTLINE: This is a dose-escalation study.

Patients receive pemetrexed disodium IV over 10 minutes and docetaxel IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced or recurrent solid tumors

  * Patients for whom docetaxel is considered appropriate anticancer therapy; docetaxel is currently approved for use in patients with the following solid tumors:

    * Non-small cell lung (NSCLC)
    * Breast
    * Prostate
    * Esophageal
    * Head and neck
    * Ovarian
    * Gastric
* Measurable or non-measurable disease
* No squamous cell NSCLC
* Controlled brain metastases allowed

  * Clinically stable with no signs of progression by MRI or CAT scan ≥ 60 days after treatment
  * Patients must be asymptomatic with no steroid requirements

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,000/mm^3*
* ANC ≥ 1,500/mm^3*
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* AST, ALT, and alkaline phosphatase (AP) must meet one of the following criteria:

  * AST or ALT ≤ 3** times upper limit of normal (ULN) AND AP normal
  * AST or ALT ≤ 1.5 times ULN AND AP ≤ 2.5 times ULN
  * AST or ALT normal AND AP ≤ 5 times ULN
* Calculated creatinine clearance ≥ 45 mL/min OR GFR measured by Tc99m-DPTA serum clearance method
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* Able to interrupt aspirin or other NSAIDs pre- and post- twice-monthly drug dosing
* Able to take folic acid, vitamin B12, or corticosteroids
* No uncontrolled serious active infections
* No pre-existing peripheral neuropathy > grade 1
* No significant cardiac disease (i.e., uncontrolled high blood pressure, unstable angina, congestive heart failure within the past 6 months, LVEF < normal, myocardial infarction within the past year, or serious cardiac arrhythmias requiring medication)
* No known severe hypersensitivity reaction to docetaxel or other drugs formulated in polysorbate 80 NOTE: *No concurrent colony-stimulating factors to maintain these values

NOTE: **For patients with liver metastases, AST or ALT ≤ 5 times ULN AND AP normal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Have received 0-1 prior systemic therapy regimens (prior adjuvant chemotherapy will be considered a prior systemic therapy regimen)
* At least 4 weeks since prior systemic anticancer therapy (6 weeks for mitomycin C and nitrosoureas)
* At least 2 weeks since prior radiotherapy and recovered from the side effects to ≤ grade 1
* At least 2 weeks since prior pleurodesis
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of combination ALIMTA and Taxotere | From first dose of the study drug until 30 days after the last administration of study medication

SECONDARY OUTCOMES:
Toxicity | From first dose of the study drug until 30 days after the last administration of study medication
Antitumor activity | From first dose of the study drug until 30 days after the last administration of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States